CLINICAL TRIAL: NCT06298006
Title: Uppföljning av Psykiatriska, Kognitiva Och Neurologiska Symtom Hos Post COVID-19 Patienter.
Brief Title: A Two Year Longitudinal Clinical Study of Neurocognitive and Psychiatric Symptoms in Post COVID-19 Patients
Acronym: PASC24
Status: Active, not recruiting | Type: Observational
Sponsor: Region Örebro County (Other)
Collaborators: Örebro University, Sweden (Other); Karolinska Institutet (Other); Karolinska University Hospital (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 275025
Record Dates: First submitted 2024-01-17; First posted 2024-03-07 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: COVID-19
Keywords: COVID-19 sequelae; cognitive symptoms; neuropsychological symptoms; neuropsychological testing; biomarkers; cerebrospinal fluid; microbiota
MeSH Terms: conditions — COVID-19; Neurobehavioral Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, cerebrospinal fluid (CSF), faeces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PASC24 study participants: Patients with residual cognitive and psychiatric symptoms after COVID-19 infection who undergo follow-up.
  Interventions: Other: Follow-up

INTERVENTIONS:
Other: Follow-up — Follow-up of neurocognitive and psychiatric symptoms in Post COVID patients (baseline, 12 months, 24 months) in correlation with biomarkers using MRI, fMRI, neuropsychological testing, lab samples (blood, CSF, microbiota).

SUMMARY:
The prospective, longitudinal, open observational study monitors patients with cognitive and neuropsychological symptoms after COVID-19 infection, in a longitudinal manner to see how the disease has affected their physical, psychological and cognitive function, their ability to be active, return to work, their health-related quality of life in correlation with potential diagnostic and prognostic markers.

DETAILED DESCRIPTION:
The aim is to increase knowledge of the underlying biological processes; how biomarkers correlate with degree of symptoms, mapping their role as diagnostic markers over time (24 months).

The investigators follow up to 100 study participants with post-acute sequelae of SARS-CoV-2 infection (PASC) for 24 months, measure their physical, psychological and neurocognitive symtoms and how they change over time (three visits: baseline, 12 months, 24 months) in correlation with biomarkers in blood, cerebrospinal fluid and faeces samples as well as neuroradiological changes on MRI (baseline, 24 months).

Knowledge about the late effects of COVID-19 and its pathogenesis is still unknown. The findings of the study can therefore be used as a guidance for future actions in healthcare and, in the best case, can lead to a possible, either curative or symptom-relieving, treatment.

ELIGIBILITY:
Inclusion Criteria:

* neurocognitive symptoms after lab-verified COVID-19 infection

Exclusion Criteria:

* severe illness e.g cancer with a short expected survival time
* ongoing alcohol abuse
* ongoing drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients:
  * who have been referred for neurocognitive symptoms after Covid-19 infection to secondary health care at Örebro University Hospital (USÖ) or who themselves sought assessment at USÖ
  * who meet inclusion criteria and do not meet exclusion criteria
  * who agreed to study participation with a written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive functions measured with Mindmore and change in cognitive profile in Mindmore. | baseline, 12 months, 24 months
  Two digital neurocognitive test batteries (Mindmore): dementia and fatigue/depression
Symptom improvement in depression | baseline, 12 months, 24 months
  Montgomery Asberg Depression Rating Scale (MADRS) has has 10 items that are completed during a clinical interview.. The items of the MADRS are as follows: apparent sadness, reported sadness inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thought, suicidal thoughts.
  MADRS assess the severity of depression. The severity of symptoms is rated by the physician. Each item has a severity scale from 0 to 6, with higher scores reflecting more severe symptoms. Ratings can be added to form an overall score (from 0 to 60) and the higher score means a worse outcome.
Self-reported symptom improvement in depression | baseline, 12 months, 24 months
  Montgomery Asberg Depression Rating Scale, Self-report version (MADRS-S) has 9-items which are based on feelings over the past 3 days. The items of the MADRS-S are as follows: Mood; Feelings of unease; Sleep; Appetite; Ability to concentrate; Initiative; Emotional involvement; Pessimism; Zest for life.
  MADRS-S assess the severity of depression. The severity of symptoms is rated by the study participant. Each item has a severity scale from 0 to 6, with higher scores reflecting more severe symptoms. Ratings can be added to form an overall score (from 0 to 54) and the higher score means a worse outcome.
Grade of self-reported mental fatigue | baseline, 12 months, 24 months
  The Mental Fatigue scale (MFS) includes 14 questions that measure mental fatigue. Questions include affective, cognitive and sensory symptoms, duration of sleep and daytime variation in symptom severity. The questions concern fatigue in general, lack of initiative, mental fatigue, mental recovery, concentration difficulties, memory problems, slowness of thinking, sensitivity to stress, increased tendency to become emotional, irritability, sensitivity to light and noise, decreased or increased sleep. One additional question includes 24-hour symptom variations. The severity of symptoms is rated by the study participant. A rating of 0 corresponds to normal function and 1-3 indicating increasing problem with the symptom (No (0), Slight (1), Fairly serious (2) and Serious (3) problems). Ratings can be added to form an overall score (from 0 to 42) and the higher score means a worse outcome.
Rate of self-reported symptoms suggestive of post-traumatic stress disorder (PTSD) | baseline, 12 months, 24 months
  The Post-traumatic Stress Disorder Checklist for The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, DSM-5 (PCL-5) is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD.
  The study partipicipant answer first a brief Criterion A för PTSD. If the answer is affirmative (i.e. PTSD is suspected) the participants continue with 20 questions (items). Each item is rated from 0 ("not at all") to 4 ("extremely") to indicate the degree to which they have been bothered by that particular symptom over the past month. Ratings can be added to form an overall score (from 0 to 80) and the higher score means a worse outcome.
Grade of self-reported stress | baseline, 12 months, 24 months
  Th Perceived Stress Scale (PSS-14) is a self-reported measure which assesses the degree to which the respondent has perceived situations in his/her life within the past month as stressful.
  The PSS-14 is comprised of 14 items intended to measure how unpredictable, uncontrollable, and overloaded individuals find their life circumstances. Individuals rate items on a 5-point Likert scale, ranging from 0 - "Never" to 4 - "Very often." Scores range from 0-56, with higher scores indicating greater perceived stress.
Grade of self-reported cognitive failures in everyday life | baseline, 12 months, 24 months
  The cognitive Failures Questionnaire (CFQ) is a self-report questionnaire consisting of 25 items assessing deficits regarding attention, perception, memory and motor functioning in everyday life. The total CFQ score is calculated by summation of all answers and scores range from 0-100. A higher total score indicates more subjective cognitive failure.

SECONDARY OUTCOMES:
Occurence of activity limitations and changes in health-related quality of life (QoL) | baseline, 12 months, 24 months
  Rating scale: the EuroQol-5 Dimension, 5 levels (EQ-5D-5L) with EuroQol-visual analogue scale (EQ-VAS)
  EQ-5D-5L assesses the current state of health in five dimensions related to well-being and function; mobility, personal care, regular activities, pain/discomfort and anxiety/depression. Each dimension has five levels from "No problems" to "extreme problems". This results in a single-digit number (from 1 to 5) that expresses the level selected for that dimension. Higher digits/scores mean en worse uotcome.
  EQ-VAS registers the patient's self-rated health in a analog scale with the minimum and maximum values: 0-100 where the endpoints are marked: 100 -"The best health you can imagine" and 0 - "The worst health you can imagine". Lower scores mean a worse outcome.
Grade of work incapacity/sick leave and time to return to work | baseline, 12 months, 24 months
  Self-assessment questionnaire.
  Study participant report grade of eventual sick-leave. According to Swedish legislation, four degrees of sick leave are possible (25%, 50%, 75%, 100%), where a higher number of percentages means worse outcome i.e. more reduced ability to work.
  They also report the time of incapacity for work (number of months of sick leave (1- 100)) where higher numbers mean worse outcome i.e. longer time of incapacity for work
Changes in body size | baseline, 12 months, 24 months
  Body mass index (BMI) gives an indication of the body size. Along with several other factors, BMI can help estimate the risk of a cardiovascular disease.
  BMI is calculated using weight and height. BMI Categories: Underweight = <18.5, Normal weight = 18.5-24.9, overweight = 25-29.9, obesity = BMI of 30 or greater. The values under 18.5 and over 25 indicate worse outcome.
Waist size | baseline, 12 months, 24 months
  The waist measurement is an indicator of the abdominal obesity that is associated with an increased risk of type 2 diabetes, cardiovascular disease and death, The values over 94cm for men and over 80cm for women indicate worse outcome i.e. abdominal obesity.
Rate of peak expiratory flow (PEF) | baseline, 12 months, 24 months
  PEF rate is the volume of air forcefully expelled from the lungs in one quick exhalation, and is an indicator of ventilation adequacy as well as airflow obstruction. Air flow is measured with the portable, hand-held device. Three readingss are performed ond the highest of three readings is used as the recorded value of the PEF Rate. PEF is measured in units of liters per minute (0-800). The expected value depends on the participant's sex, age, and height but higher numbers in the given study participant mean better outcome i.e. better lung function.
Grade of physical exercise capacity | baseline, 12 months, 24 months
  60 Second Sit-to-Stand Test (60STS) gives a measure of exercise capacity. The participant is encouraged to complete as many full stands as possible within 60 seconds. The number of full stands is registered (0-100) where higher numbers mean better outcome i.e. better physical fitness.
Concetration of Beta-Amyloid 42 in cerebrospinal fluid (CSF) as a CSF biomarker of neurodegeneration. | baseline, 24 months
  Beta-amyloid 40 and 42 are formed from amyloid precursor protein (APP) and are normally transported to the cerebrospinal fluid (CSF). In Alzheimer's disease, Beta-amyloid 42 accumulates in senile plaque and thus the level falls in CSF. Slightly lower levels of beta-amyloid 42 can also be seen in other dementia diseases.
  Cerebrospinal fluid will be collected by trained physician and results will be reported as ng/L. The expected value depends on the participant's age, but lower values in the given study participant mean worse outcome i.e. more possible neurodegeneration.
Beta Amyloid Ratio 42/40 in cerebrospinal fluid (CSF) as a CSF biomarker of neurodegeneration linked to Alzheimer's disease | baseline, 24 months
  Beta amyloid 40 is the most common variant of beta amyloid in CSF, while beta amyloid 42 predominates in senile plaques . Decreased ratio of Beta amyloid 42/40 is a strong marker of Alzheimer's disease and can be detected early in the disease progression, even before clinical dementia occurs.
  Cerebrospinal fluid will be collected by trained physician and the result is reported as a ratio. Reference interval: > 0.72 ( > 50 years of age). Lower ratio means worse outcome i.e. possible Alzheimer's disease.
Concentration of neurogranin in cerebrospinal fluid (CSF) as a CSF biomarker of neurodegeneration linked to Alzheimer's disease | baseline, 24 months
  Neurogranin is a protein expressed in synapses of the pyramidal cells of the hippocampus and cortex. Neurogranin is elevated in cerebrospinal fluid from individuals with Alzheimer's disease, but not from healthy individuals or individuals with other neurodegenerative diseases.
  Cerebrospinal fluid will be collected by trained physician and results will be reported as ng/L. The expected value depends on the participant's age, but higher values in the given study participant mean worse outcome i.e. more possible neurodegeneration.
Concentration of Tau (P-Tau) protein in cerebrospinal fluid (CSF) as a CSF biomarker of cortikal damage/neurodegeneration | baseline, 24 months
  Tau protein is a recognized biomarker of cortical damage and is assumed to be a nonspecific marker of neurodegeneration.
  Cerebrospinal fluid will be collected by trained physician and results will be reported as ng/L. The expected value depends on the participant's age, but higher values in the given study participant mean worse outcome i.e. more possible cortical damage/neurodegeneration.
Concentration of phosphorylated Tau (P-Tau) in cerebrospinal fluid (CSF) as a CSF biomarker of neurodegeneration/taupathy | baseline, 24 months
  Under physiological conditions, tau protein regulates the assembly and maintenance of the structural stability of microtubules in nerve cells. In certain brain diseases tau proteine becomes abnormally hyperphosphorylated, which ultimately causes the microtubules to disassemble, and the free tau molecules aggregate into paired helical filaments.
  Phosphorylated tau (P-tau) is assumed to be a relatively specific marker for Alzheimers disease because neurofibrillary tangles that är found in AD patients primarily consist of tau protein in the abnormally hyperphosphorylated state
  Cerebrospinal fluid will be collected by trained physician and results will be reported as ng/L. The expected value depends on the participant's age, but higher values in the given study participant mean worse outcome i.e. more possible neurodegeneration.
Concentration of neurofilament light (NFL) in cerebrospinal fluid (CSF) as a CSF biomarker of neurodegeneration | baseline, 24 months
  Neurofilament light (NFL) is a recognized biomarker of subcortical large-caliber axonal degeneration and is assumed to be a nonspecific marker of neurodegeneration.
  Cerebrospinal fluid will be collected by trained physician and results will be reported as ng/L. The expected value depends on the participant's age, but higher values in the given study participant mean worse outcome i.e. more possible neurodegeneration.
Concentration of neurofilament light (NFL) in plasma as a blood biomarker of neurodegeneration | baseline, 24 months
  Blood-based biomarkers of neurodegeneration have obvious advantages over both CSF and neuroimaging biomarkers. The collection of blood is inexpensive, noninvasive, and a more feasible measure for use in the general population, especially if serial collection is needed. Neurofilament light (NFL) is a recognized biomarker of subcortical large-caliber axonal degeneration and is assumed to be a nonspecific marker of neurodegeneration.
  Plasma will be collected by trained personnel and results will be reported as ng/L. The expected value depends on the participant's age, but higher values in the given study participant mean worse outcome i.e. more possible neurodegeneration. The values will be also compared with NFL values in cerebrospinal fluid (outcome 20), which are still the "golden standard" of NFL measurement
Occurence of APOE4 allele as biomarker of genetic predisposition to Alzheimer's disease and susceptibility to more severe course of COVID-19 infection | baseline
  The human APOE gene exists as three polymorphic alleles-ε2, ε3 and ε4-which have a worldwide frequency of 8.4%, 77.9% and 13.7%, respectively. However, the frequency of the ε4 allele is dramatically increased to ~40% in patients with late onset Alzheimers disease. APOE4 allele has also been correlated with severe COVID-19 outcomes.
  Plasma will be collected by trained personnel and results will be reported as combination of two alleles with six possible alternatives: 2/2, 2/3, 2/4, 3/3, 3/4, 4/4. Alternatives with the APOE4 allele indicate worse outcomes and combinationen: 4/4 indicates the worst possible outcome.
Brain volumes and signal abnormalities in white and gray matter | baseline, 24 months
  Imaging of the brain using Magnetic Resonance Imaging (MRI) scans. The scans are compared over time to assess changes of brain volume and progress/regression of signal abnormalities/lesions in gray and white matter
Changes in functional and structural brain connectivity | baseline, 24 months
  Imaging of the brain activity at rest using resting-state functional Magnetic Resonance Imaging (rs-fMRI). Rs-fMRI measures spontaneous low-frequency fluctuations in the BOLD signal to investigate the functional architecture of the brain and to identify various resting-state networks (RSN). The scans are compared over time to detect changes in functional and structural connectivity of the brain.
Changes in gut microbiome | Baseline, 24 months
  The gut microbiome in COVID-19 is characterized by increased fecal fungal load and increased beta-diversity (more heterogeneous), and it is unstable over time and also persistently altered after disease resolution. Assessment of gut microbiome as well as changes over time will be carried out via analysis of the fecal samples for microbial composition using 16S microbiome analysis, metabolomics and Next Generation Sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Freund-Levi, MD, PhD, Principal Investigator — Medical Faculty, Örebro University, Dept of Geriatrics, USÖ
Locations (1):
- Department of Geriatrics, University Hospital Örebro, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van den Hurk W, Bergman I, Machado A, Bjermo J, Gustavsson A. Swedish Normative Data for Mindmore: A Comprehensive Cognitive Screening Battery, Both Digital and Self-Administrated. J Int Neuropsychol Soc. 2022 Feb;28(2):188-202. doi: 10.1017/S135561772100045X. Epub 2021 May 24. PMID 34027854
- See also: Information about the study on Örebro University's website — https://www.oru.se/forskning/forskningsproj/mv/pasc/